CLINICAL TRIAL: NCT02309827
Title: A Phase 1, Randomized, Double Blind, Third-party Open, Placebo-controlled, Single And Multiple Dose Escalation, Parallel Group Study To Evaluate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Pf-06651600 In Healthy Subjects
Brief Title: Safety and Pharmacokinetic Study of PF-06651600 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: B7981001; 2014-004326-17 (EudraCT Number); PF-06651600 (Other: Alias Study Number); JAK3 (Other: Alias Study Number)
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: Inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — PF-06651600

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Cohort 1: PF-06651600 or Placebo (Experimental): Single ascending doses of PF-06651600 or placebo to evaluate safety, tolerability and PK.
  Interventions: Drug: PF-06651600 or Placebo
- Cohort 2: PF-06651600 or Placebo (Experimental): Single ascending doses of PF-06651600 or placebo to evaluate safety, tolerability and PK.
  Interventions: Drug: PF-06651600 or Placebo
- Cohort 3: PF-06651600 or Placebo (Experimental): Single ascending doses and multiple ascending doses of PF-06651600 or placebo to evaluate safety, tolerability and PK.
  Interventions: Drug: PF-06651600 or Placebo
- Cohort 4: PF-06651600 or Placebo (Experimental): Single ascending doses and multiple ascending doses of PF-06651600 or placebo to evaluate safety, tolerability and PK.
  Interventions: Drug: PF-06651600 or Placebo
- Cohort 5: PF-06651600 or Placebo (Experimental): Single ascending doses and multiple ascending doses of PF-06651600 or placebo to evaluate safety, tolerability and PK.
  Interventions: Drug: PF-06651600 or Placebo
- Cohort 6: PF-06651600 or Placebo (Experimental): Single ascending doses and multiple ascending doses of PF-06651600 or placebo to evaluate safety, tolerability and PK.
  Interventions: Drug: PF-06651600 or Placebo
- Cohort 7: PF-06651600 or Placebo (Experimental): Single ascending doses and multiple ascending doses of PF-06651600 or placebo to evaluate safety, tolerability and PK.
  Interventions: Drug: PF-06651600 or Placebo
- Cohort 8: PF-06651600 or Placebo (Experimental): Single ascending doses and multiple ascending doses of PF-06651600 or placebo to evaluate safety, tolerability and PK.
  Interventions: Drug: PF-06651600 or Placebo
- Cohort 9: PF-06651600 or Placebo (Experimental): Multiple ascending doses of PF-06651600 or placebo to evaluate safety, tolerability and PK.
  Interventions: Drug: PF-06651600 or Placebo

INTERVENTIONS:
Drug: PF-06651600 or Placebo — PF-06651600 or placebo will be administered as an extemporaneously prepared solution in each cohort.

SUMMARY:
This study is a first in human study of PF-06651600. PF-06651600 is being developed for treatment of inflammatory bowel disease. This study will test single and multiple doses of PF-06651600. The goal of the study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of PF-06651600 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male/female subjects between 18 and 55 years old, inclusive. Females must be of non-child bearing potential.
* BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Evidence of personally signed and dated informed consent document.
* Willing and able to comply with scheduled visits, treatment plan, lab tests and other study procedures.
* Subjects must avoid high intensity UV light exposure (eg, active sunbathing, tanning beds/booths or sunlamps) from the first dose of study drug and for the duration of the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, GI, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Use of tobacco/nicotine containing products in excess of 5 cigarettes/day.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males.
* Screening blood pressure >140/90 mm Hg.
* Screening laboratory abnormalities as defined by the protocol.
* Unwilling or unable to comply with the Lifestyle Guidelines as defined by the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
24 hour creatinine clearance (Single Dose) | Single dose period, Day 0 (baseline) and 24 hours post dose Day 1.
  24 hour urine creatinine clearance in healthy subjects participating in the single dose periods. For the single dose period, assessment occurs on Study Days 0 and 1.
24 hour creatinine clearance (Multiple Dose) | Multiple dose period, Days 0 (baseline), 7 and 14.
  24 hour urine creatinine clearance in healthy subjects participating in the multiple dose period. For the multiple ascending dose period assessments occur on Study Days 7 and 14.
Change from baseline in urine volume (Single Dose) | Single dose period, Day 0 (baseline) and 24 hours post dose Day 1.
  For the single dose period, assessment occurs on Study Days 0 and 1.
Change from baseline in urine electrolytes (Single Dose) | Single dose period, Day 0 (baseline) and 24 hours post dose Day 1.
  For the single dose period, assessment occurs on Study Days 0 and 1.
Change from baseline in urine osmolality (Single Dose) | Single dose period, Day 0 (baseline) and 24 hours post dose Day 1.
  For the single dose period, assessment occurs on Study Days 0 and 1.
Change from baseline of urine volume (Multiple Dose) | Multiple dose period, Days 0 (baseline), 7 and 14.
  For the multiple ascending dose period assessments occur on Study Days 7 and 14.
Change from baseline of urine electrolytes (Multiple Dose) | Multiple dose period, Days 0 (baseline), 7 and 14.
  For the multiple ascending dose period assessments occur on Study Days 7 and 14.
Change from baseline in urine osmolality (Multiple Dose) | Multiple dose period, Days 0 (baseline), 7 and 14.
  For the multiple ascending dose period assessments occur on Study Days 7 and 14.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) for PF-06651600 (Single Dose) | 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Maximum Observed Plasma Concentration (Cmax)
Maximum Observed Plasma Concentration (Cmax) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Maximum Observed Plasma Concentration (Cmax)
Time to Reach Maximum Observed Plasma Concentration (Cmax) for PF-06651600 (Single Dose) | 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Time to Reach Maximum Observed Plasma Concentration (Cmax)
Time to Reach Maximum Observed Plasma Concentration (Cmax) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Time to Reach Maximum Observed Plasma Concentration (Cmax)
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for PF-06651600 (Single Dose) | 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf)
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06651600 (Single Dose) | 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Dose Normalized Maximum Observed Plasma Concentration (Cmaxdn) for PF-06651600 (Single Dose) | 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Dose Normalized Maximum Observed Plasma Concentration (Cmaxdn)
Dose Normalized Maximum Observed Plasma Concentration (Cmaxdn) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Dose Normalized Maximum Observed Plasma Concentration (Cmaxdn)
Dose Normalized Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinfdn) for PF-06651600 (Single Dose) | 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Dose Normalized Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinfdn)
Dose Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClastdn) for PF-06651600 (Single Dose) | 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Dose Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClastdn)
Plasma Decay Half-Life (t1/2) for PF-06651600 (Single Dose) | 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Plasma Decay Half-Life (t1/2)
Plasma Decay Half-Life (t1/2) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Plasma Decay Half-Life (t1/2)
Mean Resonance Time (MRT) for PF-06651600 (Single Dose) | 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Mean Resonance Time (MRT)
Mean Resonance Time (MRT) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Mean Resonance Time (MRT)
Apparent Volume of Distribution (Vz/F) for PF-06651600 (Single Dose) | 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Apparent Volume of Distribution (Vz/F) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Apparent Total Body Clearance (CL/F) for PF-06651600 (Single Dose) | 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent total body clearance (CL/F) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Total Body Clearance (CL/F) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent total body clearance (CL/F) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Minimum Observed Plasma Concentration (Cmin) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Minimum Observed Plasma Concentration (Cmin)
Average Concentration for Dosing Interval (12 or 24 hours) (Cav) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Average Concentration for Dosing Interval (12 or 24 hours) (Cav)
Area Under the Curve for Dosing Interval (12 or 24 hours) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Area Under the Curve for Dosing Interval (12 or 24 hours)
Dose Normalized Area Under the Curve for Dosing Interval (12 or 24 hours) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Dose Normalized Area Under the Curve for Dosing Interval (12 or 24 hours)
Peak to Trough Fluctuation (PTF) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Peak to Trough Fluctuation (PTF)
Observed Accumulation Ratio (Rac) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Observed Accumulation Ratio (Rac)
Observed Accumulation Ratio for Cmax (RacCmax) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Observed Accumulation Ratio for Cmax (RacCmax)
Steady State Accumulation Ratio (Rss) for PF-06651600 (Multiple Dose) | Days 1, 4, 6, 8, 10, 12 and 14 (0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48 hours post dose)
  Steady State Accumulation Ratio (Rss)
Amount of PF-066561600 Excreted Unchanged (Multiple Dose) | Day 14 (12, 24 hours post dose)
  Concentration in urine.
Change from baseline of BCL2 gene expression in whole blood (Single Dose) | Days -1 and 1 (0, 1, 2, 4, 8, 12 and 24 hours post dose)
Change from baseline of BCL2 gene expression in whole blood (Multiple Dose) | Days 1, 5, 10, 14 (0, 1, 2, 4, 8, 12 and 24 hours post dose), 16, and 28
Change from baseline of IP-10 protein concentration in serum (Multiple Dose) | Days 0, 2, 7, 14 (0, and 16 hours post dose) and 16
Change from baseline of hsCRP protein concentration in serum (Multiple Dose) | Days 0, 2, 7, 14 (0, and 16 hours post dose) and 16
Change from baseline of reticulocyte counts in whole blood (Single Dose) | Days 0, 2, 3, and 7
Change from baseline of neutrophil counts in whole blood (Single Dose) | Days 0, 2, 3, and 7
Change from baseline of hemoglobin level whole blood (Single Dose) | Days 0, 2, 3, and 7
Change from baseline of reticulocyte counts in whole blood (Multiple Dose) | Days 0, 4, 8, 12, 14 (pre-dose) 15, and 28
Change from baseline of neutrophil counts in whole blood (Multiple Dose) | Days 0, 4, 8, 12, 14 (pre-dose) 15, and 28
Change from baseline of hemoglobin level in whole blood (Multiple Dose) | Days 0, 4, 8, 12, 14 (pre-dose) 15, and 28
Renal Clearance (Multiple Dose) | Day 1, Day 14 (12, 24 hours post dose)
Percentage of PF-066561600 Excreted Unchanged (Multiple Dose) | Day 14 (12, 24 hours post dose)
  Concentration in urine.
Change from baseline of IP-10 gene expression in blood (Multiple Dose) | Days 0, 5, 10, 14 (0, 1, 2, 4, 8 and 12 hours post dose) and 16
Change from baseline of IP-10 gene expression in blood (Single Dose) | Days 0, 1 (0, 1, 2, 4, 8 and 12 hours post dose) and 16

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- [Derived] Saadeddin A, Purohit V, Huh Y, Wong M, Maulny A, Dowty ME, Sagawa K. Virtual Bioequivalence Assessment of Ritlecitinib Capsules with Incorporation of Observed Clinical Variability Using a Physiologically Based Pharmacokinetic Model. AAPS J. 2024 Jan 24;26(1):17. doi: 10.1208/s12248-024-00888-9. PMID 38267790
- [Derived] Wojciechowski J, S Purohit V, Huh Y, Banfield C, Nicholas T. Evolution of Ritlecitinib Population Pharmacokinetic Models During Clinical Drug Development. Clin Pharmacokinet. 2023 Dec;62(12):1765-1779. doi: 10.1007/s40262-023-01318-3. Epub 2023 Nov 2. PMID 37917289
- [Derived] Purohit V, Huh Y, Wojciechowski J, Plotka A, Salts S, Antinew J, Dimitrova A, Nicholas T. Leveraging Prior Healthy Participant Pharmacokinetic Data to Evaluate the Impact of Renal and Hepatic Impairment on Ritlecitinib Pharmacokinetics. AAPS J. 2023 Mar 28;25(3):32. doi: 10.1208/s12248-023-00792-8. PMID 36977960
- [Derived] Telliez JB, Dowty ME, Wang L, Jussif J, Lin T, Li L, Moy E, Balbo P, Li W, Zhao Y, Crouse K, Dickinson C, Symanowicz P, Hegen M, Banker ME, Vincent F, Unwalla R, Liang S, Gilbert AM, Brown MF, Hayward M, Montgomery J, Yang X, Bauman J, Trujillo JI, Casimiro-Garcia A, Vajdos FF, Leung L, Geoghegan KF, Quazi A, Xuan D, Jones L, Hett E, Wright K, Clark JD, Thorarensen A. Discovery of a JAK3-Selective Inhibitor: Functional Differentiation of JAK3-Selective Inhibition over pan-JAK or JAK1-Selective Inhibition. ACS Chem Biol. 2016 Dec 16;11(12):3442-3451. doi: 10.1021/acschembio.6b00677. Epub 2016 Nov 10. PMID 27791347
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7981001